CLINICAL TRIAL: NCT04542850
Title: An Open-Label, Pilot Study to Evaluate the Safety, Tolerability, and Efficacy of 5-Aminolevulinic Acid Phosphate and Sodium Ferrous Citrate (5-ALA-Phosphate + SFC) in Subjects With SARS-CoV-2 Infection (COVID-19)
Brief Title: Pilot Study to Evaluate the Safety, Tolerability, and Efficacy of 5-ALA-Phosphate + SFC in Subjects With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons in Ireland - Medical University of Bahrain (Other)
Collaborators: Bahrain Defence Force Hospital (Other); Salmaniya Medical Complex (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68 / 02-Aug-2020
Record Dates: First submitted 2020-08-16; First posted 2020-09-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV 2; COVID-19
Keywords: 5-ALAPhosphate + SFC; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Sodium Glutamate

STUDY DESIGN:
Intervention Model Description: This is an open label pilot study involving 40 patients with COVID-19 disease. Patients that are hospitalized due to confirmed SARS-CoV-2 infection will be assigned to two groups according o their severity grade (moderate or severe).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moderate group and Severe Group (Other): Moderate group and Severe group - . Both groups will be administered 5-aminolevulinic acid (5-ALA) is a natural delta amino acid widely present in nature that can be found in common food. 5-ALA combined with sodium ferrous citrate (SFC) produces the nutritional dietary supplement 5-ALA-Phosphate + SFC (5-ALA + SFC).
  Interventions: Dietary Supplement: 5-ALA-Phosphate + SFC (5-ALA + SFC)

INTERVENTIONS:
Dietary Supplement: 5-ALA-Phosphate + SFC (5-ALA + SFC) — Moderately ill hospitalized patients will receive:
  250 mg 5-ALA-Phosphate and 143.4 mg SFC (15.2 mg as Fe) two times daily (resulting in 500 mg 5-ALA-Phosphate and 286.8 mg SFC (30.4 mg as Fe) daily) for 7 days, then 250 mg 5-ALA-Phosphate and 143.4 mg SFC (15.2 mg as Fe) once daily for 21 days
  Severely ill hospitalized patients will receive:
  250 mg 5-ALA-Phosphate and 143.4 mg SFC (15.2 mg as Fe) three times daily (resulting in 750 mg 5-ALA-Phosphate and 430.2 mg SFC (45.6 mg as Fe) daily) for 7 days, then 250 mg 5-ALA-Phosphate and 143.4 mg SFC (15.2 mg as Fe) once daily for 21 days

SUMMARY:
This is an open-label, interventional exploratory study to evaluate the safety and efficacy of 5-ALA-Phosphate + SFC in subjects with acute moderate or severe respiratory illness secondary to infection with SARS-CoV-2 virus (COVID-19) involving 40 subjects.

The primary objective is to evaluate the safety of 4-week oral administration of 5-ALAPhosphate + SFC. This study is expected to last for 4 weeks and will include follow-up until day 28 in the hospital or in an outpatient setting if the subjects are discharged earlier.

DETAILED DESCRIPTION:
This is an open-label, interventional exploratory study to evaluate the safety and efficacy of 5-ALA-Phosphate + SFC in subjects with acute moderate or severe respiratory illness secondary to infection with SARS-CoV-2 virus (COVID-19).

Heme is critical for appropriate oxygen binding and delivery to remote site and without the heme contained within the hemoglobin tetramer, multicellular organisms would be unable to survive. Furthermore HO-1 degrades heme into biliverdin, carbon monoxide (CO), and iron, and biliverdin is immediately reduced and turned into bilirubin by biliverdin reductase. Biliverdin/bilirubin and CO both have anti-oxidative functions and they regulate important biological processes like inflammation, apoptosis, cell proliferation, fibrosis, and angiogenesis. Therefore, HO-1 is deemed to be a promising drug target (Ryter 2006). HO-1 is a major anti-inflammatory enzyme and a key regulator that induces immune tolerance. 5-ALA-Phosphate + SFC increases heme metabolism and HO-1 via enhancement of porphyrin biology and utilizes the HO-1 for endothelial pacification strategy.

The primary endpoints of this study is- all treatment emergent AEs and SAEs Grade III and IV (CTC) with reasonable possibility of causal relationship to 5-ALA-Phosphate + SFC. 40 subjects with symptoms requiring hospitalization will be enrolled in thestudy, with 20 subjects enrolled in each group below:

Group 1: 20 Moderately ill hospitalized subjects not requiring assisted ventilation Group 2: 20 Severely ill hospitalized subjects requiring assisted ventilation

The duration of this clinical study will be 4 weeks, and follow-up will be performed until Day 28 in hospital, or in an outpatient setting if subjects improve and are discharged home or to alternative care facility.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent, or with a legal representative who can provide informed consent
2. Aged ≥ 21 to 70 years
3. Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection confirmed by polymerase chain reaction (PCR) test before beginning study dose regime
4. qSOFA ≥ 1
5. Currently hospitalized
6. Moderate COVID-19 patients should meet any of the following criteria:

   evidence of lower respiratory disease by clinical assessment (qSOFA ≥ 1or imaging) and saturation of oxygen (SpO2) ≥94% on room air at sea level.

   Severe COVID-19 patients should meet any of the following criteria: a respiratory frequency >30 breaths per minute, SpO2 <94% on room air at sea level, ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mmHg, and lung infiltrates >50% (if possible to measure). In exceptional cases the investigator can decide due to certain signs and symptoms to assign a moderate patient to the severe group although not all criteria mentioned before are fulfilled (to be documented with explanation).
7. Radiographic evidence (chest X-ray or chest CT scan) of pulmonary infiltrates
8. Able to swallow 5 capsules of study product at dosing time points.

Exclusion Criteria:

1. Subject has critical symptoms of COVID19 infection as defined as: high-flow oxygen therapy (>15 l/min delivered by nasal cannula or mask) or invasive mechanical ventilation signifying respiratory failure, septic shock, and/or multiple organ dysfunction ventilation at screening.
2. Subject is nourished via a nasogastric tube
3. Subject has acute or chronic type(s) of porphyria or a family history of porphyria
4. Subject has demonstrated previous intolerance of 5-ALA and/or SFC by topical or oral administration (except for photosensitivity)
5. Pregnant or nursing women
6. Males and females of reproductive potential who have not agreed to use an
7. adequate method of contraception during the study For females, adequate birth control methods will be defined as: hormonal contraceptives, intrauterine device or double barrier contraception, i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam For males, adequate birth control methods will be defined as double barrier contraception, i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam For females, menopause is defined as one year without menses; if in question, a folliclestimulating hormone of >40 U/ml must be documented. Hysterectomy, bilateral oophorectomy,or bilateral tubal ligation must be documented, as applicable
8. Subjects who are unable or unwilling to comply with requirements of the clinical trial
9. Participation in any other clinical trial of an experimental treatment for COVID-19
10. Evidence of multiorgan failure
11. Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 X upper limit of normal (ULN)
12. Creatinine clearance < 50 mL/min using the Cockcroft-Gault formula for participants ≥ 18 years of age {Cockcroft 1976}
13. Any other reason that makes the subject unsuitable in the Investigator's opinion

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
The incidence of treatment emergent Adverse Events (safety and tolerability) of 5-ALA-Phospate + SFC in patients with acute moderate or severe respiratory illness secondary to infection with SARS-CoV-2 virus (COVID-19). | 28 days
  To describe the incidence of treatment-emergent Adverse Events (TEAEs) of CTC Grades III and IV within four weeks following base line dose.

SECONDARY OUTCOMES:
Sum COVID-19 Modified Ordinal Scale for Clinical Improvement maximum daily score over 28 days of dosing for Moderate group and for Severe group | 28 days
  To describe patient's condition in Moderate and Severe group using average, median, minimum and maximum in COVID-19 Modified Ordinal Scale for Clinical Improvement score.
Rate of change in COVID-19 Modified Ordinal Scale for Clinical Improvement maximum daily score over 28 days of dosing for individual subjects in Moderate group and in Severe group | 28 days
  To describe patient´s condition in Moderate and Severe Group using rate of change in COVID-19 Modified Ordinal Scale for Clinical Improvement score.
Patient and subgroup profile of COVID-19 Modified Ordinal Scale for Clinical Improvement score vs. days hospitalized | 28 days
  To describe patient´s condition in Moderate and Severe Group using patient and subgroup profile of COVID-19 Modified Ordinal Scale for Clinical Improvement score vs. days hospitalized.
Overall survival | day 14 and day 28
  To describe time until death from any cause
Results of investigator´s assessment of patient´s oxygen therapy | 28 days
  To describe patient´s blood oxygenation
Results of mechanical ventilation settings | 28 days
  To describe mechanical ventilation settings course during study.
Results of duration of ventilation | from date of enrolment until the extubation or until last 5-ALA- Phosphate -SFC administration on day 28
  To describe duration of patient´s ventilation
The time to resolution of patient´s symptoms | 28 days
  To describe patient´s specific symptoms course during study.
Results of patient´s oxygen saturation (respiratory parameters) | 28 days
  To describe patient´s oxygen saturation course during study.
Length of hospitalization | From date of enrolment until last 5-ALA- Phosphate -SFC administration at day 28
  To describe duration of hospitalization in the patient groups.
The total time in ICU | From date of enrolment until last 5-ALA- Phosphate -SFC administration at day 28
  To describe duration of residence in ICU in the patient groups.
Results of investigator´s assessment of patient´s condition using (q)SOFA score | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe patient´s (q)SOFA score course during study.
Results of patient´s PT parameter | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe patient´s coagulation function course during study which by evaluating the PT value.
Results of patient´s D-Dimer parameter | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe patient´s coagulation function course during study which by evaluating the D-Dimer value.
Results of patient´s PTT parameter | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe patient´s coagulation function course during study which by evaluating the PTT value.
Results of patient´s SARS-CoV-2 viral load status (efficacy) | day 7, 14 and 28
  To describe patient's SARS-CoV-2 viral load course during study.
Results of patient´s Procalcitonin level. | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe infection parameter course of each patient during study by evaluating the Procalcitonin value.
Results of patient´s IL-6 level | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe infection parameter course of each patient during study by evaluating the IL-6 value.
Results of patient´s Serum Ferritin level | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe infection parameter course of each patient during study by evaluating the Serum ferritin value.
Results of patient´s C-Reactive protein (CRP) level | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe infection parameter course of each patient during study by evaluating the C-Reactive protein (CRP) value.
Results of patient´s T helper cells (CD4/CD8) level. | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe infection parameter course of each patient during study by evaluating the T helper cells (CD4/CD8) value.
Results of patient´s Bilirubin level. | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe infection parameter course of each patient during study by evaluating the Bilirubin value.
Results on patient´s Leucocytes | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Leucocytes value
Results on patient´s Neutrophils | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Neutrophils value
Results on patient´s Lymphocyte | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Lymphocyte value
Results on patient´s Platelets | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Platelets value
Results on patient´s Hemoglobin | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Hemoglobin value
Results on patient´s Albumin | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Albumin value
Results on patient´s AST | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating AST value
Results on patient´s ALT | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating ALT value
Results on patient´s Total bilirubin | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Total bilirubin value
Results on patient´s Blood urea nitrogen | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Blood urea nitrogen value
Results on patient´s Serum creatinine | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Serum creatinine value
Results on patient´s Creatinine kinase | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Creatinine kinase value
Results on patient´s LDH | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating LDH value
Results on patient´s Myoglobin glucose | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating Myoglobin glucose value
Results on patient´s aPTT | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating aPTT value
Results on patient´s urine | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating urinalysis (urine test strip)
Results on hepatic function | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating hepatic function
Results on patient´s renal function | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating renal function
Results on patient´s iron parameters | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe laboratory assessments course during study by evaluating iron parameters
Results on patient´s physical examination | day 0, 2, 3, 5, 7, 10, 14, 21, 28
  To describe patient´s conditions course during study using physical examination which include General Appearance, ENT, Respiratory, Cardiovascular, Musculoskeletal, Skin and Neurological.
Results on patient´s Co-infections | 28 days
  To describe patient's Co-infections course during study.
Results on patient´s Care Level | 28 days
  To describe patient´s care level course during study.
Results on patient´s Mean arterial pressure(MAP) | 28 days
  To describe patient´s vital signs course during study by evaluating Mean arterial pressure(MAP)
Results on patient´s heart rate (HR) | 28 days
  To describe patient´s vital signs course during study by evaluating heart rate (HR)
Results on patient´s respiratory rate (RR) | 28 days
  To describe patient´s vital signs course during study by evaluating respiratory rate (RR)
Results on patient´s 12-lead ECG | day 0, 7, 14 and 28
  To describe patient´s 12-lead ECG result course during study.
Organ damage | 28 days
  To describe patient´s organ damage status during the study

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Darwish, Dr, Principal Investigator — Bahrain Defense Force Royal Medical Services, Military Hospital
Locations (2):
- Bahrain (2):
  - Bahrain Defense Force Royal Medical Services, Military Hospital, Manama
  - Salmaniya Medical Complex, Manama

IPD SHARING:
Plan to Share IPD: Yes
Monitoring, audits, and REC review will be permitted and provide direct access to source data and documents. The Lead PI and the researchers assigned by him will have access to the stored data/specimens. Only the Lead PI and the researchers assigned working on this study will be eligible to obtain the data/specimens from the participants during data collection.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be collected in the case report form to allow for cross referencing to check validity.
  Study documents (paper) will be retained in a secure (kept locked when not in use) location during and after the trial has finished. All essential documents including source documents will be retained for a period of 5 years after study completion (last patient, last study point).
Access Criteria: Study documents (paper) will be retained in a secure (kept locked when not in use) location during and after the trial has finished.

REFERENCES:
- [Background] El Kalamouni C, Frumence E, Bos S, Turpin J, Nativel B, Harrabi W, Wilkinson DA, Meilhac O, Gadea G, Despres P, Krejbich-Trotot P, Viranaicken W. Subversion of the Heme Oxygenase-1 Antiviral Activity by Zika Virus. Viruses. 2018 Dec 20;11(1):2. doi: 10.3390/v11010002. PMID 30577437
- [Background] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Background] Devadas K, Dhawan S. Hemin activation ameliorates HIV-1 infection via heme oxygenase-1 induction. J Immunol. 2006 Apr 1;176(7):4252-7. doi: 10.4049/jimmunol.176.7.4252. PMID 16547262
- [Background] Hill-Batorski L, Halfmann P, Neumann G, Kawaoka Y. The cytoprotective enzyme heme oxygenase-1 suppresses Ebola virus replication. J Virol. 2013 Dec;87(24):13795-802. doi: 10.1128/JVI.02422-13. Epub 2013 Oct 9. PMID 24109237
- [Background] Hooper PL. COVID-19 and heme oxygenase: novel insight into the disease and potential therapies. Cell Stress Chaperones. 2020 Sep;25(5):707-710. doi: 10.1007/s12192-020-01126-9. Epub 2020 Jun 4. PMID 32500379
- [Background] Ibanez FJ, Farias MA, Retamal-Diaz A, Espinoza JA, Kalergis AM, Gonzalez PA. Pharmacological Induction of Heme Oxygenase-1 Impairs Nuclear Accumulation of Herpes Simplex Virus Capsids upon Infection. Front Microbiol. 2017 Oct 31;8:2108. doi: 10.3389/fmicb.2017.02108. eCollection 2017. PMID 29163402
- [Background] Ito H, Nishio Y, Hara T, Sugihara H, Tanaka T, Li XK. Oral administration of 5-aminolevulinic acid induces heme oxygenase-1 expression in peripheral blood mononuclear cells of healthy human subjects in combination with ferrous iron. Eur J Pharmacol. 2018 Aug 15;833:25-33. doi: 10.1016/j.ejphar.2018.05.009. Epub 2018 May 10. PMID 29753693
- [Background] Nishio Y, Fujino M, Zhao M, Ishii T, Ishizuka M, Ito H, Takahashi K, Abe F, Nakajima M, Tanaka T, Taketani S, Nagahara Y, Li XK. 5-Aminolevulinic acid combined with ferrous iron enhances the expression of heme oxygenase-1. Int Immunopharmacol. 2014 Apr;19(2):300-7. doi: 10.1016/j.intimp.2014.02.003. Epub 2014 Feb 13. PMID 24530569
- [Background] Ogawa K, Sun J, Taketani S, Nakajima O, Nishitani C, Sassa S, Hayashi N, Yamamoto M, Shibahara S, Fujita H, Igarashi K. Heme mediates derepression of Maf recognition element through direct binding to transcription repressor Bach1. EMBO J. 2001 Jun 1;20(11):2835-43. doi: 10.1093/emboj/20.11.2835. PMID 11387216
- [Background] Protzer U, Seyfried S, Quasdorff M, Sass G, Svorcova M, Webb D, Bohne F, Hosel M, Schirmacher P, Tiegs G. Antiviral activity and hepatoprotection by heme oxygenase-1 in hepatitis B virus infection. Gastroenterology. 2007 Oct;133(4):1156-65. doi: 10.1053/j.gastro.2007.07.021. Epub 2007 Jul 25. PMID 17919491
- [Background] Ryter SW, Alam J, Choi AM. Heme oxygenase-1/carbon monoxide: from basic science to therapeutic applications. Physiol Rev. 2006 Apr;86(2):583-650. doi: 10.1152/physrev.00011.2005. PMID 16601269
- [Background] Saito K, Fujiwara T, Ota U, Hatta S, Ichikawa S, Kobayashi M, Okitsu Y, Fukuhara N, Onishi Y, Ishizuka M, Tanaka T, Harigae H. Dynamics of absorption, metabolism, and excretion of 5-aminolevulinic acid in human intestinal Caco-2 cells. Biochem Biophys Rep. 2017 Jul 13;11:105-111. doi: 10.1016/j.bbrep.2017.07.006. eCollection 2017 Sep. PMID 28955775
- [Background] Schmidt WN, Mathahs MM, Zhu Z. Heme and HO-1 Inhibition of HCV, HBV, and HIV. Front Pharmacol. 2012 Oct 4;3:129. doi: 10.3389/fphar.2012.00129. eCollection 2012. PMID 23060790
- [Background] Tseng CK, Lin CK, Wu YH, Chen YH, Chen WC, Young KC, Lee JC. Human heme oxygenase 1 is a potential host cell factor against dengue virus replication. Sci Rep. 2016 Aug 24;6:32176. doi: 10.1038/srep32176. PMID 27553177
- [Background] Zhong M, Wang H, Ma L, Yan H, Wu S, Gu Z, Li Y. DMO-CAP inhibits influenza virus replication by activating heme oxygenase-1-mediated IFN response. Virol J. 2019 Feb 20;16(1):21. doi: 10.1186/s12985-019-1125-9. PMID 30786886
- [Background] Brooks A., Study 8259980 5-ALA/SFC: A Phase I, Double-Blind, Placebo-Controlled, Single and Multiple Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Caucasian and Japanese Subjects, Covance: Leeds and London, UK (2013)
- [Background] Investigator's Brochure, SBI Pharmaceuticals Internal Document: 5-Aminolevulinic Acid (5-ALA)Phosphate Version 1.0. July, 2020
- [Background] Matsumoto C., Study ALA-01 "Bioequivalence study of test foods A, B, and C - Based on the PlasmaConcentration of 5-Aminolevulinic Acid." Kaiyu Clinic: Tokyo Japan (2010)
- [Background] World Health Organization (WHO) R&D Blueprint: Novel Coronavirus COVID-19 Therapuetic Trial Synopsis. Draft dated February 18, 2020. Accesssed online 09Jul20 at https://www.who.int/blueprint/priority-diseases/key-action/COVID- 19_Treatment_Trial_Design_Master_Protocol_synopsis_Final_18022020.pdf